CLINICAL TRIAL: NCT05462002
Title: Intrinsic Foot Muscle Morphology and Function in Runners With and Without Plantar Fasciitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lau On Yue, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: PF_IFM_Training
Record Dates: First submitted 2022-07-08; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fascitis
Keywords: intrinsic foot muscle, plantar fasciitis, runners, balance, postural control
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- plantar fasciitis group: Distance runners with plantar fasciitis
- asymptomatic control group: Distance runners without plantar fasciitis

SUMMARY:
Plantar fasciitis is one of the most common musculoskeletal conditions in distance runners. 44% of patients still had the symptoms after 15 years from the first onset. The chronicity of the condition may lead to significant limitations on daily activities and even cessation of running. In the concept of foot core system, the intrinsic foot muscles work together with plantar fascia to stabilize the foot arches and provide dynamic support to the foot during functional activities. Given that the intrinsic foot muscles also play an important role as a direct sensors of foot deformation, postural control may be compromised during pathological state. Therefore, this study aim to investigate the differences in the muscle thickness and cross-sectional area of intrinsic foot muscles and postural control in runners with and without plantar fasciitis. We hypothesized that runners with plantar fasciitis demonstrate small intrinsic foot muscles sizes and poor postural control when compared with the asymptomatic counterparts.

DETAILED DESCRIPTION:
this is a case-control study, using ultrasound imaging (USG) to examine the differences in muscle thickness (MT) and cross-sectional area (CSA) of Abductor Hallucis (AbH), flexor hallucis brevis (FHB), flexor digitorum brevis (FDB), and quadratus plantae (QP), and postural control in runners with and without plantar fasciitis. All participants were recruited through recruitment flyers and word of mouth from local running community. The dependent variables included navicular height using navicular drop test, foot posture using the 6-item Foot Posture Index (FPI-6). The actual status of symptoms was evaluated by visual analog scale (VAS) pain at the first steps in the morning, VAS pain at worst of the day, the Foot Function Index Revised short form (FFI-R S), and the Foot and Ankle Ability Measure (FAAM).

The postural control was assessed by three 10-seconds eyes opened trials and three 10-seconds eyes closed trials single-leg stance recorded on an instrumented force platform . (AMTI. Watertown, MA) at 50 Hz. Center of pressure velocity (cm/s) was calculated for each condition using Balance Clinic software (AMTI. Watertown, MA). In addition, percent modulation was calculated using equation 1 to provide an estimate of a participant's reliance on visual information for the postural control of intrinsic foot muscles.

Equation 1 is as followed.

% modulation= (eyes open velocity-eyes closed velocity)/(eyes open velocity)

Larger negative values represent a greater impairment to postural control when vision is removed and suggest a greater reliance on visual information.

ELIGIBILITY:
Inclusion Criteria:

* distance runners who run more than 20km per week for at least 2 years. Runners who were between 18 and 60 years of age with symptoms of chronic plantar fasciitis: if they reported tenderness on palpation of the medial calcaneal tuberosity, thickness of plantar fascia >4.0mm at insertion with USG, and exhibited one of the following complaints: 1. plantar heel pain > 1 month; 2 pain on the first step in the morning or after prolonged sitting; 3. pain on prolonged standing; 4 pain when running.

Exclusion Criteria:

* Those who had undergone surgery to the plantar fascia, or had local injection within the last 3 months, or had any coexisting painful musculoskeletal condition of the lower limb, or any neurological or systematic disease were excluded

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: distance runners who run more than 20km per week for at least 2 years.
Sampling Method: Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Muscle thickness (MT) of Abductor Hallucis (AbH), Flexor Hallucis Brevis (FHB), Flexor Digitorum Brevis (FDB), Quadratus Plantae (QP) | baseline
  ultrasound measurement
Cross sectional area (CSA) of Abductor Hallucis (AbH), Flexor Hallucis Brevis (FHB), Flexor Digitorum Brevis (FDB), Quadratus Plantae (QP) | baseline
  ultrasound measurement
postural control | baseline
  three 10-seconds eyes opened trials and three 10-seconds eyes closed trials single-leg stance recorded on an instrumented force platform. percent modulation was calculated using equation 1 to provide an estimate of a participant's reliance on visual information for the postural control of intrinsic foot muscles.
  Equation 1 is as followed.
  % modulation= (eyes open velocity-eyes closed velocity)/(eyes open velocity)
  Larger negative values represent a greater impairment to postural control when vision is removed and suggest a greater reliance on visual information.
Visual Analog Scale (VAS) pain at first steps in the morning | baseline
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Visual Analog Scale (VAS) worst pain of the day | baseline
  measuring 100 mm in length marked from 0 (absence of pain) to 100 mm (worst imaginable pain)
Foot and Ankle Ability Measure (FAAM) | baseline
  Higher scores represent higher levels of function, with 100% representing no dysfunction.
Foot Function Index revised short form (FFI-RS) | baseline
  grade 1 corresponds to no pain and 4 corresponds to worst pain imaginable. The numerical 5 is not used as a score but is used to indicate that the subscale question is not applicable for the participant. Higher scores represent higher levels of pain, stiffness, difficulty, activity limitation, and psychosocial aspect

SECONDARY OUTCOMES:
Foot posture index (FPI) | Baseline
  Pronated postures are given a positive value, the higher the value the more pronated.
Navicular drop | Baseline
  Supinated foot (<5mm); Neutral foot (5-9mm); pronated foot (>9mm)

CONTACTS AND LOCATIONS:
Overall Officials: On Yue Lau, PhD candidate, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- CUHK-ORT Sports Injury Research Laboratory, Shatin, Hong Kong